CLINICAL TRIAL: NCT01292681
Title: Multi-modality Imaging in the Prediction of Response to Systemic Treatment in Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MICC
Record Dates: First submitted 2011-02-01; First posted 2011-02-09 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; FDG-PET-CT; MRS,; DCE-MRI; DWI; colorectal cancer with histologically proven distant metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multi-modality imaging (Other)
  Interventions: Other: Multi-modality imaging

INTERVENTIONS:
Other: Multi-modality imaging — Week -2-0 FDG-PET-CT,1H MRS, DCE-MRI, DWI Week 1 1H MRS, DCE-MRI, DWI, 19F MRS, FDG-PET-CT Week 9 FDG-PET-CT

SUMMARY:
Because of metastatic liver cancer of the colon or rectum, patients will be treated with cytotoxic drugs (chemotherapy). In the Radboud University Nijmegen Medical Centre the investigators investigate whether the imaging techniques at an early stage of treatment can predict which patients will have benefited from this treatment.

In the study the investigators use two different scanners: a MR (magnetic resonance) scanner and a PET (Positron Emission Tomography) scanner combined with a CT (Computer Tomography) scanner. An MR scanner is a large magnet and looks like a CT scanner which also makes pictures. But instead of using X-rays the recordings are made with magnetic fields. The scan consists of a table on which the patient will lie with the head in a half-dome with a camera. The examination with the MR scan is not painful and not harmful.

The PET scan is a type of CT scan that makes (after administration of a radioactive liquid), a scan of (part of) the body. The amount of radioactivity that is used for the study is so small that it will not have an adverse impact on the patient. This research is two times combined with a''normal''CT scan.

Using the MR scan, the investigators can research the oxygensupply, the aggressiveness of the tumour and the degree of liver metastases that die from the chemotherapy . The investigators can also, after administration of a MR contrast agent, investigate the blood supply of a tumor through imaging. If you are treated with the chemotherapeutic drug capecitabine the investigators can monitor the intake of this agent in the liver metastases. The PET CT scan tells us more about the metabolism in the liver metastases.

DETAILED DESCRIPTION:
Colorectal cancer is a frequently occurring cancer and about half of the patients develop distant metastases to the liver. Only a subset of patients respond to systemic treatment, which is potentially toxic and expensive. Therefore, predictive markers are needed to determine treatment efficacy at an early stage. Preferably, they should provide insight into the biology of colorectal cancer liver metastasis. In the past it has been shown that several biomarkers as assessed with PET, MRI and MRS can serve as predictive markers. Response to systemic therapy depends on several factors: delivery of the drug by the tumor vascular system; cellular uptake, retention and metabolism; intrinsic sensitivity to a specific drug. The relative contribution of these factors to response will be different for different drugs. Since systemic treatment of colorectal cancer involves a combination of drugs, predictive markers should be sensitive to a range of these factors. In this project we propose the integrated analysis of noninvasive functional and molecular in vivo imaging methods in order to predict the response to treatment in patients with liver metastases of colorectal cancer. Tumor vascularity can be assessed by dynamic contrast enhanced magnetic resonance imaging (DCE-MRI). The fluoropyrimidines FU and capecitabine - which are part of standard treatment regimens - contain a fluorine atom which can be measured by fluorine-19 MR spectroscopy (19F MRS). The intracellular uptake and metabolism of drugs is an energy-consuming process. 18F-Fluoro-2-deoxyglucose positron emission tomography (FDG-PET) provides information on glucose uptake and hexokinase activity. Tumor characterization in terms of grade and aggressiveness may give a relevant approximation to the intrinsic sensitivity of a tumor to a drug. With 1H MRS the total amount of choline (tCho), a precursor of cell membranes, can be measured. Tumor cellularity and extracellular matrix composition can be assessed with diffusion weighted MRI (DWI).

The aim of this study is to obtain data on the biology data of colorectal cancer liver metastasis, namely tumor vascularization (DCE-MRI), tumor cellularity (DWI), tumor (choline) metabolism (1H MRS) and tumor glucose metabolism (FDG-PET). These data will be correlated with the clinical outcome of patients and with drug uptake and metabolism (19F MRS). We will study the relative contribution of each imaging method to predict the outcome of patients with colorectal cancer at an early stage.

Research questions:

1. Do pre-treatment characteristics of liver metastases of colorectal cancer as assessed by dynamic contrast enhanced MRI (DCE-MRI), diffusion weighted MRI (DWI), 1H MR spectroscopy (MRS) and FDG-PET predict treatment outcome?
2. Do early changes (one week after start of treatment) in DCE-MRI, DWI, 1H MRS and FDG-PET characteristics of liver metastases of colorectal cancer predict treatment outcome?
3. Do 19F MRS parameters of fluoropyrimidine metabolism in liver metastases of colorectal cancer predict treatment outcome at an early stage (one week after start of treatment)?
4. What is the relative contribution of each above mentioned imaging method to predict treatment outcome of colorectal liver metastases? Design: 60 patients with liver metastases of colorectal cancer treated with fluoropyrimidine-based therapy will participate to the study. Baseline 1H MRS of the liver will be performed in a session at 3 Tesla followed by DCE-MRI and DWI at 1.5 Tesla. FDG-PET will be added to the standard baseline CT scan, using our clinical PET-CT scanner. DCE-MRI, DWI, 1H and 19F MRS as well as FDG-PET of the liver will be repeated one week after start of treatment. Clinical response will be evaluated after three treatment cycles by FDG-PET-CT. We will assess the relative contribution of each imaging method as well as the integrated use of these methods for the identification of predictive biomarkers for response to treatment.

Relevance of this study: Since the response of a tumor to systemic drugs may be highly variable between patients, a method that predicts the sensitivity of a tumor to treatment at an early stage would enable individualization of therapy and consequently would protect patients against the toxic effects of ineffective treatment. Preferably, those predictive markers should also give us further insight into the biology of colorectal cancer. For this reason we propose to study a combination of in vivo noninvasive imaging methods which allow the monitoring of relevant biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Histological proven colorectal cancer with histologically proven distant metastases.
* First line fluoropyrimidine-based treatment for liver metastases of colorectal cancer containing fluoropyrimidines.
* Measurable liver metastases of at least 2 cm.
* Age minimal 18 years.
* Written informed consent

Exclusion Criteria:

* Prior chemotherapy within six months before start of the study.
* Contra-indication for MR and/or PET examinations (e.g. pacemaker, claustrophobia, diabetes mellitus).
* Karnofsky Performance Status <70.
* Diffuse liver metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Correlation early changes in imaging and treatment outcome | imaging before start, week 1, week 9
  Correlation early changes in imaging and treatment outcome Week -2-0: PET-CT and MRI Week 0 Start chemotherapy Week 1 PET-CT and MRI Week 9 PET-CT onderzoek

SECONDARY OUTCOMES:
Correlation pretreatment imaging values and treatment outcome | imaging before start, week 1 and week 9
  Correlation pretreatment imaging values and treatment outcome Week -2-0: PET-CT and MRI Week 0 Start chemotherapy Week 1 PET-CT and MRI Week 9 PET-CT onderzoek

CONTACTS AND LOCATIONS:
Overall Officials: C.J.A. Punt, Md PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands